CLINICAL TRIAL: NCT01593358
Title: Venous Obstruction in Neurodegenerative Disorders Research Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Synergy Health Concepts, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RESEARCH_REGISTRY
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Cerebral Spinal Venous Insufficiency
Keywords: CCSVI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To establish if there are venous obstructions in patients with neurodegenerative disorders

DETAILED DESCRIPTION:
This research registry will observe the venous obstruction in neurodegenerative disorders. This will provide data that will allow researchers to classify abnormal valve and venous morphology, distinguish vessels which are more responsive to treatment, determine groups who respond more favorably to treatment, and overall evaluate the outcomes of venous angioplasty in various neurodegenerative disorders that involve venous obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the nature of the study, including the risks and benefits and execute an informed consent
* Males or Females between the ages of 18 and 90 years of age
* Voluntary agreement to participate in the Venous Obstructions in Neurodegenerative Diseases Research Registry

Exclusion Criteria:

* Any implantable/metallic objects that prevent subject from having a magnetic resonance imaging ( MRI/MRV) study
* History of uncontrolled hypertension
* Previous venous angioplasty treatment for Chronic cerebral spinal venous insufficiency
* Special Populations. Special groups include, but are not limited to children, prisoners, pregnant women,fetuses, and cognitively impaired individuals who are unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human subjects will be approached for participation in this registry that are receiving or seeking medical care at Synergy Health Concepts, Inc.No individuals shall be excluded from participation in the Research Registry based on race, ethnicity, or gender.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08; Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph Hewett, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Synergy Health Concepts, Inc., Newport Beach, California, United States